CLINICAL TRIAL: NCT03412318
Title: Evaluation of the Effect of Root Canal Preparation by TF and M-Pro on Post-Operative Pain After Single Visit Endodontic Treatment: A Blinded Randomized Clinical Trial Therapeutic Study.
Brief Title: Evaluation of the Effect of Root Canal Preparation by TF and M-Pro on Post-Operative Pain After Single Visit Endodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmad Abdul Aziz Almorad, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TF vs Mpro
Record Dates: First submitted 2018-01-08; First posted 2018-01-26 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Acute Pulpitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Twisted file (Experimental): Use of twisted file during cleaning and shaping of root canals
  Interventions: Device: Twisted file
- Mpro (Active Comparator): Use of Mpro file during cleaning and shaping of root canals
  Interventions: Device: Mpro

INTERVENTIONS:
Device: Twisted file — Use of twisted file during cleaning and shaping of root canals
  Arms: Twisted file
Device: Mpro — Use of Mpro during cleaning and shaping of root canals
  Arms: Mpro

SUMMARY:
A study to comparatively evaluate the post operative pain between root canal preparation by reciprocating file (TF) and full rotation file (M-Pro) in patients with single rooted teeth with acute irreversible pulpits.

DETAILED DESCRIPTION:
Teeth with symptomatic irreversible pulpitis are selected according to the eligibility and exclusion criteria and patients are then randomized to receive treatment after using Twisted files or M-pro files. The treatment is done in single visit. The postoperative pain is then assessed using the Numerical Rating Scale 6,12, 24 and 48 hours post-instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good health (American Society of Anesthesiologists Class II or higher).
* Patients having symptomatic irreversible pulpitis in their single rooted teeth.
* Age range is between 20 and 60 years.
* Patients who can understand numerical rating scale (NRS).
* Patients able to sign informed consent.

Exclusion Criteria:

* Patients with positive percussion test.
* Patients having history of necrosis with or without apical pathosis.
* Patients have sinus tract or fistula extra oral or intraoral.
* Pregnant or mentally retarded patients.
* Teeth with grade 2 or 3 mobility.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-06 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 2 days
  Post-operative pain assessed after treatment using the NRS pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad Almorad, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gambarini G, Testarelli L, De Luca M, Milana V, Plotino G, Grande NM, Rubini AG, Al Sudani D, Sannino G. The influence of three different instrumentation techniques on the incidence of postoperative pain after endodontic treatment. Ann Stomatol (Roma). 2013 Mar 20;4(1):152-5. doi: 10.11138/ads.0152. Print 2013 Jan. PMID 23741536